CLINICAL TRIAL: NCT05625373
Title: The Effect of Intrawound Vancomycin Powder on Surgical Site Infection in Inguinal Lymph Node Dissection
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Jessica DiSilvestro, Principle Investigator, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1895541
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 unblinded to either receive vancomycin powder in the operating room or no vancomycin powder (no placebo utilized).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vancomycin powder (Experimental): Women randomized to receive vancomycin powder will receive 1g into each of the irrigated inguinal surgical beds (maximum of 2g dose per patient). After dissection and irrigation of the surgical bed, the operating room staff will open the medication vial and sterilely dispense the medication into a sterile container. The surgeon will place the medication powder into the irrigated and hemostatic surgical bed. The procedure will be repeated on the opposite side after dissection.
  Interventions: Drug: Vancomycin
- No vancomycin powder (No Intervention): Patient randomized to the no vancomycin arm will not receive the intraoperative antibiotic. Their surgery will follow standard protocol. No placebo will be utilized.

INTERVENTIONS:
Drug: Vancomycin — The powder will be placed within the surgical wound prior to skin closure.
  Arms: Vancomycin powder

SUMMARY:
The study will be a pilot randomized control trial with a 1:1 patient randomization of vancomycin powder placement at the time of surgery (compared to no vancomycin placement) with the goal of reducing postoperative complications in patients undergoing an inguinal lymph node dissection for vulvar cancer. The primary objective is to measure the composite rate of postoperative complications within 30 days of inguinal lymph node dissection in patients with vulvar cancer.

DETAILED DESCRIPTION:
The aim of the study is to investigate the impact of intrawound vancomycin powder on surgical site infections. The primary objective is to measure the composite rate of postoperative complications, including inguinal wound infection (superficial and deep surgical site infection), inguinal incision separation, and hospital readmission within 30 days of inguinal lymph node dissection in women with vulvar cancer.

Secondary objectives include assessing the rate of seroma or lymphocele development within 30 days of surgery. Adverse events including allergic reactions (systemic or local hypersensitivity reactions) and antibiotic resistant infections (based on wound cultures) will be described.

The study will be a pilot randomized control trial with a 1:1 patient randomization of vancomycin powder placement at the time of surgery. The investigators will identify women who are planning to undergo inguinal lymph node dissection for vulvar cancer and after consented will be randomized to either receive intrawound vancomycin powder in the operating room or to not receive intrawound vancomycin powder. Women randomized to receive vancomycin powder will receive 1g into each of the irrigated inguinal surgical beds (maximum of 2g dose per patient).

Patients will be followed post operatively at their standard postoperative visits typically at 1-3 week intervals until adequate healing of their incisions. An electronic questionnaire will be administered to all patients at the postoperative visits between 3-6 weeks to assess recovery and complications. Outcomes will be collected until six weeks postoperatively. The study will be conducted at a single institution

ELIGIBILITY:
Inclusion Criteria:

* Women who are undergoing inguinal lymph node dissection for vulvar dysplasia
* Women with a prior lymph node dissection >30 days before
* Women undergoing either a sentinel lymph node biopsy or full lymphadenectomy in a unilateral or bilateral groin dissection

Exclusion Criteria:

* Known allergy to vancomycin
* Known resistance to vancomycin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2024-04-25 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Composite rate of postoperative complications | Within 30 days after surgery
  Rate of composite postoperative complications including inguinal wound infection (superficial and deep surgical site infection), inguinal incision separation, and hospital readmission within 30 days

SECONDARY OUTCOMES:
Antibiotic resistant infections | Within 30 days after surgery
  Rate of antibiotic resistant infections based on wound cultures of a postoperative infection
Allergic reactions | Within 30 days after surgery
  Rate of systemic or local hypersensitivity reactions of the inguinal incision

CONTACTS AND LOCATIONS:
Overall Officials: Jessica DiSilvestro, MD, Principal Investigator — Women & Infants Hospital
Locations (1):
- Women and Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DiSilvestro JB, Zitek E, Robison K, Ebott J, Jansen C, Eurich K, Mathews C, DiSilvestro P, Oliver M, Stuckey A, Miller K, Lokich E. The effect of intrawound vancomycin powder on surgical site infection in inguinal lymph node dissection: a randomized controlled trial pilot study. Gynecol Oncol Rep. 2025 May 9;59:101765. doi: 10.1016/j.gore.2025.101765. eCollection 2025 Jun. PMID 40487852